CLINICAL TRIAL: NCT05201209
Title: LASER FiLaC™ (FISTULA LASER CLOSURE) : First-line Treatment of Complex Anal Fistulas
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: LASER FILAC 2
Record Dates: First submitted 2019-08-01; First posted 2022-01-21 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2019-08

CONDITIONS: Complex Anal Fistula
Keywords: Fistula; Laser; Sphincter
MeSH Terms: conditions — Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Complex anal fistula is a fistula whose treatment with fistulotomy would expose the patient to an excessive risk of post-operative continence disorders. It is a challenge in proctological surgery because of the complexity of its therapeutic management in relation to the recurrences' frequency and the need to preserve sphincter function. Indeed, management is mainly based on fistulotomy techniques, but the latter expose patients to a significant alteration of their continence (less than 10% incontinence for simple fistulas but 30-50% for complex fistulas). In addition, these fistulas' management is constraining for patients due to the need for multiple interventions, long-term post-operative care and repeated discontinuation of activity.

Sphincteral saving techniques have therefore developed over the last three decades and have enriched the therapeutic panel of complex fistulas. They aim to block fistula pathways without risking altering sphincter function. In addition, their surgical consequences are often simple. However, they are associated with a greater risk of failure than after fistulotomy and sometimes disappointing to the point that some of these techniques have been gradually abandoned (biological glue and plug for example).

Among these sphincteral saving techniques, the investigators know the advancement flap, the injection of biological glue, plug's installation, the LIFT (Ligation of Inter sphincteric Fistula Tract), the clip's use but also, more recently a laser treatment, FiLaC™ (for Fistula Laser Closure), knowing that the idea was not new since the ND-YAG3 and CO24.5 lasers were already used in the treatment of anal fistulas, about twenty years ago, in experimental studies.

This technique consists of radiating 360° laser energy radially into the fistula path to "burn" it and causing thermal destruction by coagulation of the fistula wall ans granulation tissue2. It can bo offered to any type of fistula at risk on continence, including horseshoe extensions that can be treated at the same time. It is well suited for outpatient management because the postoperative period is simple and painless.

The literature is still poor on the subject with some studies published openly but the preliminary results are encouraging with a success rate of about 70%. No continence disorders reported.

DETAILED DESCRIPTION:
A first retrospective study was conducted in the medical and surgical proctology department of the Hospital Group Paris Saint-Joseph on a cohort on 69 consecutive patients seen between May 2016 ans April 2017 and treated by FiLaC™ for a complex anal fistula. This technique has thus cured 60% of patients with superior trans-sphincter fistula. No incontinence-type complications were observed. These results, all the interesting as it was a learning phase, led the investigators to continue to use FiLaC™, which is currently practiced by all the team's practitioners as a first-line sphincter savings technique. The idea of this new work is to conduct an evaluation on a larger cohort of patients now that the investigators have more experience and it is being used routinely in the department at Groupe Hospitalier Paris Saint-Joseph.

ELIGIBILITY:
Inclusion Criteria:

* Patient with complex anal fistula treated by the FiLaC™ between 05/01/17 and 05/01/18

Exclusion Criteria:

* Patient scheduled for treatment by FiLaC™ and collected as such but finally treated by fistulotomy given a fistula pathway considered intraoperatively less complex than expected
* Patient with recto vaginal or vaginal skin fistula
* Patient under guardianship or curators
* Patient deprived of liberty
* Patient objecting to the use of their data for this research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with complex anal fistula treated by the FiLaC™ between 05/01/17 and 05/01/18
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2019-06-02 (Actual); Study Completion 2019-06-02 (Actual)

PRIMARY OUTCOMES:
Assess on a larger scale the cure rate of patients treated by the proctology department between May 2017 and May 2018 for complex anal fistula. | 6 months
  Clinical cure rate (in percentage) of complex anal fistula treated with FiLaC at the last medical contact in Groupe Hospitalier Paris Saint-Joseph.

SECONDARY OUTCOMES:
Identify predictive factors for clinical fistula healing to determine the best indications. | 6 months
  This outcome corresponds to evaluate the correlations between patients' clinical characteristics and cure rates.
Confirm on a larger scale the absence of anal incontinence after treatment with FiLaC™ . | 1 year
  Comparison of Wexner's scores before and after the intervention. This score evaluates the importance of anal incontinence, it varies from 0 to 20, 20 corresponding to total incontinence.
  It is criticized for varying too much according to the transit.
Description of possible complications | 1 year
  This outcome corresponds to the number of events per person of other complications after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Vincent De PARADES, M.D, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

REFERENCES:
- [Background] Limura E, Giordano P. Modern management of anal fistula. World J Gastroenterol. 2015 Jan 7;21(1):12-20. doi: 10.3748/wjg.v21.i1.12. PMID 25574077
- [Background] Wilhelm A. A new technique for sphincter-preserving anal fistula repair using a novel radial emitting laser probe. Tech Coloproctol. 2011 Dec;15(4):445-9. doi: 10.1007/s10151-011-0726-0. Epub 2011 Aug 16. PMID 21845480
- [Background] Ellison GW, Bellah JR, Stubbs WP, Van Gilder J. Treatment of perianal fistulas with ND:YAG laser--results in twenty cases. Vet Surg. 1995 Mar-Apr;24(2):140-7. doi: 10.1111/j.1532-950x.1995.tb01308.x. PMID 7778253
- [Background] Bodzin JH. Laser ablation of complex perianal fistulas preserves continence and is a rectum-sparing alternative in Crohn's disease patients. Am Surg. 1998 Jul;64(7):627-31; discussion 632. PMID 9655272
- [Background] Slutzki S, Abramsohn R, Bogokowsky H. Carbon dioxide laser in the treatment of high anal fistula. Am J Surg. 1981 Mar;141(3):395-6. doi: 10.1016/0002-9610(81)90207-5. PMID 6782904
- [Background] Giamundo P, Geraci M, Tibaldi L, Valente M. Closure of fistula-in-ano with laser--FiLaC: an effective novel sphincter-saving procedure for complex disease. Colorectal Dis. 2014 Feb;16(2):110-5. doi: 10.1111/codi.12440. PMID 24119103
- [Background] Dudukgian H, Abcarian H. Why do we have so much trouble treating anal fistula? World J Gastroenterol. 2011 Jul 28;17(28):3292-6. doi: 10.3748/wjg.v17.i28.3292. PMID 21876616
- [Background] Soltani A, Kaiser AM. Endorectal advancement flap for cryptoglandular or Crohn's fistula-in-ano. Dis Colon Rectum. 2010 Apr;53(4):486-95. doi: 10.1007/DCR.0b013e3181ce8b01. PMID 20305451
- [Background] Lindsey I, Smilgin-Humphreys MM, Cunningham C, Mortensen NJ, George BD. A randomized, controlled trial of fibrin glue vs. conventional treatment for anal fistula. Dis Colon Rectum. 2002 Dec;45(12):1608-15. doi: 10.1007/s10350-004-7247-0. PMID 12473883
- [Background] Swinscoe MT, Ventakasubramaniam AK, Jayne DG. Fibrin glue for fistula-in-ano: the evidence reviewed. Tech Coloproctol. 2005 Jul;9(2):89-94. doi: 10.1007/s10151-005-0204-7. Epub 2005 Jul 8. PMID 16007368
- [Background] Johnson EK, Gaw JU, Armstrong DN. Efficacy of anal fistula plug vs. fibrin glue in closure of anorectal fistulas. Dis Colon Rectum. 2006 Mar;49(3):371-6. doi: 10.1007/s10350-005-0288-1. PMID 16421664
- [Background] Ortiz H, Marzo J, Ciga MA, Oteiza F, Armendariz P, de Miguel M. Randomized clinical trial of anal fistula plug versus endorectal advancement flap for the treatment of high cryptoglandular fistula in ano. Br J Surg. 2009 Jun;96(6):608-12. doi: 10.1002/bjs.6613. PMID 19402190
- [Background] Ozturk E, Gulcu B. Laser ablation of fistula tract: a sphincter-preserving method for treating fistula-in-ano. Dis Colon Rectum. 2014 Mar;57(3):360-4. doi: 10.1097/DCR.0000000000000067. PMID 24509460
- [Background] Rojanasakul A, Pattanaarun J, Sahakitrungruang C, Tantiphlachiva K. Total anal sphincter saving technique for fistula-in-ano; the ligation of intersphincteric fistula tract. J Med Assoc Thai. 2007 Mar;90(3):581-6. PMID 17427539
- [Background] Liu WY, Aboulian A, Kaji AH, Kumar RR. Long-term results of ligation of intersphincteric fistula tract (LIFT) for fistula-in-ano. Dis Colon Rectum. 2013 Mar;56(3):343-7. doi: 10.1097/DCR.0b013e318278164c. PMID 23392149
- [Background] Herreros MD, Garcia-Arranz M, Guadalajara H, De-La-Quintana P, Garcia-Olmo D; FATT Collaborative Group. Autologous expanded adipose-derived stem cells for the treatment of complex cryptoglandular perianal fistulas: a phase III randomized clinical trial (FATT 1: fistula Advanced Therapy Trial 1) and long-term evaluation. Dis Colon Rectum. 2012 Jul;55(7):762-72. doi: 10.1097/DCR.0b013e318255364a. PMID 22706128
- [Background] Giamundo P, Esercizio L, Geraci M, Tibaldi L, Valente M. Fistula-tract Laser Closure (FiLaC): long-term results and new operative strategies. Tech Coloproctol. 2015 Aug;19(8):449-53. doi: 10.1007/s10151-015-1282-9. Epub 2015 Feb 28. PMID 25724967